CLINICAL TRIAL: NCT04824170
Title: Effects of Neural Glides Versus Proprioceptive Neuromuscular Facilitation in Terms of Joint Position Sense and Pain in Cervical Radiculopathy
Brief Title: Effects of Neural Glides Versus Proprioceptive Neuromuscular Facilitation in Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/19/2031 Ayesha Niaz
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural glide (Experimental): Neural mobilization of median nerve which includes gliding and sliding was given
  Interventions: Other: Neural Glide
- Rhythmic stabilization technique (Experimental): Proprioceptive Neuromuscular Facilitation (Rhythmic stabilization technique will be Given)
  Interventions: Other: Rhythmic stabilization technique

INTERVENTIONS:
Other: Neural Glide — hot pack and cervical traction is applied for 10-15 min.Group A received Neural mobilization of median nerve which includes gliding and sliding was given,therapist stood on the patient & affected side besides the patient, patient'S shoulder was depressed with one hand and elbow was moved in 90 degree flexion, forearm supination, extend the wrist and fingers with other hand. Then patient arm was moved into 90 degree abduction and then sliding or gliding of nerve was applied. Sliding was applied with elbow extension and wrist flexion and elbow flexion with wrist extension. 6 sets were performed. Each set was performed for 60 seconds, for alternative days in week for 4 weeks and then progressed to gliding/tensioning technique when symptoms improved
  Arms: Neural glide
Other: Rhythmic stabilization technique — This group was receiving (PNF) Rhythmic stabilization technique with base line treatment.
  Subject was lying in spine position on the treatment table and therapist resist an isometric contraction of agonist muscle group.pt maintain this position for 10 sec without trying to move and 12-15 repetitions were performed with 30 sec rest. Each therapeutic session treatment was focused on facilitation of neck stabilizers, improving neck stability, coordination, decreasing pain and improving postural control
  Arms: Rhythmic stabilization technique

SUMMARY:
this project was a Quasi-Experimental Trial. conducted to compare the Effects of Neural Glides Versus Proprioceptive Neuromuscular Facilitation in Terms of Joint Position Sense and Pain in Cervical Radiculopathy . so that we can have best treatment option for patients with cervical radiculopathy

DETAILED DESCRIPTION:
non probability convenient sampling was done. patients following eligibility criteria from Madina Teaching Hospital FSD and Kadijatulkubra hospital Chiniot. Non Probability Convenient sampling was done. Sample size was calculated with G power. 28 Participants were randomly allocated in two groups equally via convenient sampling method. Baseline assessment was done initially. Group A was given neural glides and Group B was given PNF along with conventional physiotherapy treatment (hot pack and traction). Duration of research was almost 6 months. Intervention was applied for 4 weeks, 3 sessions per week. Pre and Post treatment readings were taken in 1st and 4th week session Assessment was done via Numeric Pain Rating Scale; NDI, CVA and JPE as subjective measurements. All participants were provided written informed consent prior to commencement of the procedures. They were free to quit the treatment at any stage of research. Data was analyzed by using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral upper extremity pain, parenthesis, or numbness.
* Neck Disability Index (NDI) score of 10/50 points or greater.
* Numeric pain rating scale scoring (moderate pain).
* Craniovertebral angle measured less than 49 with forward head posture.
* Positive distraction test, Upper limb tension test, spurling test.

Exclusion Criteria:

* Any red flags (tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis etc.
* Central nervous system involvement.
* History of whiplash injury within the previous 6weeks.
* Prior surgery to the cervical or thoracic spine from 6 months ago.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
pain by numeric pain rating scale | 2 months
  0-10 , 0 minimum 10 maximum pain
Functional disability by NECK DISABILITY INDEX | 2 months
  This means that the overall score range is between 0 and 50, 0 being no to little pain and discomfort while 50 being the severest degree of pain and disability with complete activity limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Niaz, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sokunbi OG, Muhwati L, Robinson P. A Randomized Controlled trials on the effects of acupuncture and proprioceptive neuromuscular facilitation (PNF) on supraspinatus tendinitis. IOSR Journal of Dental and Medical Sciences. 2014;13(11):63-9.